CLINICAL TRIAL: NCT05098756
Title: The Effectiveness of Applying Art Therapy on Social Interaction, Self-esteem and Well-Being for Elderly Residents in Long-Term Care Institutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Tsui-Wei Chien, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C110024
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Long-Term Care; Aged
Keywords: Elderly Residents; Long-Term Care Institutions; Social Interaction; Self-esteem; Well- Being; Art Therapy
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art therapy group (Experimental): Experimental group received 8-week art therapy. Art therapy uses different themes and materials to art-making.
  Interventions: Other: Art therapy
- No intervention group (No Intervention): No intervention group maintain the institution's original daily routine and participation in activities.

INTERVENTIONS:
Other: Art therapy — The art therapy in this study is once a week, 90 minutes each section for a total of 8-week, and using theme-oriented group art therapy. Each section has one theme, and the researcher guides the elderly to make artistic creations. Each section includes a warm-up phase is 15 minutes, the creative phase is 60 minutes, and sharing phase is 15 minutes.
  Arms: Art therapy group

SUMMARY:
When aging, older people migrate to long-term care institutions. The elderly residents lack autonomy due to the characteristics of group life. The decline of health function or the occurrence of diseases can easily lead to reduced physical activity, decreased interpersonal interaction, social withdrawal, low self-esteem, and decreased well-being. In current that emphasizes the elderly in health promotion and disease prevention activities, art therapy can be applied for the elderly to achieve the purpose of health promotion. Art therapy could effectively improve social interaction, self-esteem, and well-being; but many researchers still suggest that it is necessary to investigate the effectiveness of art therapy for elderly residents in long-term care institutions. The purpose of this study is to explore the effectiveness of art therapy in improving social interaction, self-esteem, and well-being for elderly residents in long-term care institutions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older and lived in the same long-term care institution for more than three months.
* Communicate in Mandarin or Taiwanese.
* With glasses or hearing aids and other assistive devices can have good vision and hearing functions.
* Both upper limb muscle power ≥ 4 points, can autonomous movement against moderate resistance. Under supervision, can safely use scissors for artistic creation and sit continuously for 90 minutes.
* Score > 20 points on Barthel Index.
* Score > 16 points on Mini-Mental Status Examination.
* Score ≤ 9 points on Geriatric Depression Scale.
* After the researcher's explanation, the participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Under 65 years of age, and lived in the same long-term care institution less than three months.
* Severe hearing and vision impaired, making it impossible to communicate.
* Receiving antidepressant drugs or related treatments.
* Completely dependent on activities of daily living.
* Severe depression or severe dementia.
* The elderly are participating in artistic creation-related activities.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Socially Supportive Activity Inventory | After 8-week art therapy
  An index-type instrument allows evaluating the quantity and quality of elders' participation in social activity in long-term care settings (Hsu, 2011). All organized into nine subcategories, including (1) all social contacts with family members and friends, (2) chatting with acquaintances, (3) holiday-related activities, (4) cognitive games, (5) involvement by outside organizations, (6) entertainment, (7) pleasure trips, (8) arts/crafts classes, and (9) religious activities (Hsu, 2011). Each subcategory contained three components: frequency, meaningfulness, and enjoyment (Hsu, 2011). The frequency ranged from 1 to 9, and meaningful-ness and enjoyment rated on a 4-point Likert rating ranged from 1 to 4 (Hsu, 2011). Higher scores represented more frequent participation in the activity, more significant meaning to one's life, and greater enjoyment in activity participation (Hsu, 2011).

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale(Chinese version) | After 8-week art therapy
  A 10-item scale measured the self-esteem of the respondent (Yeung, 1998). All items answered on a 4-point Likert rating, the minimum and maximum scores on the scale are 10 and 40, with lower scores suggesting better self-esteem (Yeung, 1998).
Well-Being Scale for Elders | After 8-week art therapy
  A 9-item scale measured the well-being of the elderly (Lien & Chen, 2015). All items answered on a 5-point Likert rating, the minimum and maximum scores on the scale are 9 and 45, with higher scores suggesting better well-being (Lien & Chen, 2015).

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Long-term care facility, New Taipei City
  - Long-term care facility, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ciasca EC, Ferreira RC, Santana CLA, Forlenza OV, Dos Santos GD, Brum PS, Nunes PV. Art therapy as an adjuvant treatment for depression in elderly women: a randomized controlled trial. Braz J Psychiatry. 2018 Jul-Sep;40(3):256-263. doi: 10.1590/1516-4446-2017-2250. Epub 2018 Feb 1. PMID 29412335
- [Result] Hsu YC. Socially supportive activity inventory: reliability and validity of a social activity instrument for long-term care institutions. J Nurs Res. 2011 Sep;19(3):161-72. doi: 10.1097/JNR.0b013e318229c479. PMID 21857323
- [Result] Karpaviciute S, Macijauskiene J. The Impact of Arts Activity on Nursing Staff Well-Being: An Intervention in the Workplace. Int J Environ Res Public Health. 2016 Apr 19;13(4):435. doi: 10.3390/ijerph13040435. PMID 27104550
- [Result] Kim H, Kim S, Choe K, Kim JS. Effects of Mandala Art Therapy on Subjective Well-being, Resilience, and Hope in Psychiatric Inpatients. Arch Psychiatr Nurs. 2018 Apr;32(2):167-173. doi: 10.1016/j.apnu.2017.08.008. Epub 2017 Aug 24. PMID 29579508
- [Result] Kinney JM, Rentz CA. Observed well-being among individuals with dementia: Memories in the Making, an art program, versus other structured activity. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):220-7. doi: 10.1177/153331750502000406. PMID 16136845
- [Result] Laranjeira C, Campos C, Bessa A, Neves G, Marques MI. Mental Health Recovery Through "Art Therapy": A Pilot Study in Portuguese Acute Inpatient Setting. Issues Ment Health Nurs. 2019 May;40(5):399-404. doi: 10.1080/01612840.2018.1563255. Epub 2019 Apr 3. PMID 30943062
- [Result] Nan JKM, Ho RTH. Effects of clay art therapy on adults outpatients with major depressive disorder: A randomized controlled trial. J Affect Disord. 2017 Aug 1;217:237-245. doi: 10.1016/j.jad.2017.04.013. Epub 2017 Apr 11. PMID 28433887
- [Result] Radl D, Vita M, Gerber N, Gracely EJ, Bradt J. The effects of Self-Book(c) art therapy on cancer-related distress in female cancer patients during active treatment: A randomized controlled trial. Psychooncology. 2018 Sep;27(9):2087-2095. doi: 10.1002/pon.4758. Epub 2018 Jun 10. PMID 29744966
- [Result] Richards AG, Tietyen AC, Jicha GA, Bardach SH, Schmitt FA, Fardo DW, Kryscio RJ, Abner EL. Visual Arts Education improves self-esteem for persons with dementia and reduces caregiver burden: A randomized controlled trial. Dementia (London). 2019 Oct-Nov;18(7-8):3130-3142. doi: 10.1177/1471301218769071. Epub 2018 Apr 13. PMID 29653492
- [Result] Roswiyani R, Kwakkenbos L, Spijker J, Witteman CLM. The Effectiveness of Combining Visual Art Activities and Physical Exercise for Older Adults on Well-Being or Quality of Life and Mood: A Scoping Review. J Appl Gerontol. 2019 Dec;38(12):1784-1804. doi: 10.1177/0733464817743332. Epub 2017 Nov 21. PMID 31640495
- [Result] Seifert K, Spottke A, Fliessbach K. Effects of sculpture based art therapy in dementia patients-A pilot study. Heliyon. 2017 Nov 22;3(11):e00460. doi: 10.1016/j.heliyon.2017.e00460. eCollection 2017 Nov. PMID 29264417
- [Result] Ching-Teng Y, Ya-Ping Y, Yu-Chia C. Positive effects of art therapy on depression and self-esteem of older adults in nursing homes. Soc Work Health Care. 2019 Mar;58(3):324-338. doi: 10.1080/00981389.2018.1564108. Epub 2019 Jan 10. PMID 30628552
- See also: Self-esteem reinforcement strategies in ADHD: comparison between hypnosis and art-therapy — https://doi.org/10.1016/j.ejpn.2017.04.1290
- See also: A randomized, controlled study of the effects of art therapy on older Korean-Americans' healthy aging — https://doi.org/10.1016/j.aip.2012.11.002
- See also: The practice of spiritual care in the long-term care facilities in Taiwan — https://doi.org/10.6317/LTC.201912_23(3).0006
- See also: The development of the well-being scale for elders in Taiwan — http://www.airitilibrary.com/Publication/alDetailedMesh?DocID=19966822-201503-201503200015-201503200015-29-37
- See also: The factors affecting the relocation adjustment for the residents: A case study of a long term care facility in Taipei — http://www.airitilibrary.com/Publication/alDetailedMesh?DocID=22195777-201312-201401030003-201401030003-19-36
- See also: The effect of integrating rational emotive behavior therapy and art therapy on self-esteem and resilience — https://doi.org/10.1016/j.aip.2012.12.006